CLINICAL TRIAL: NCT02376543
Title: Comparison Study in Pancreatic Fiducial Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped for change in needle usage
Sponsor: Parkview Health (Other)
Responsible Party: Principal Investigator, Neil Sharma, M.D., Interventional Gastroenterologist, Parkview Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRC14-1020 Pancreatic Fiducial
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 19 Gauge EUS FNA BNX (Active Comparator): Subjects receiving EUS and fluoroscopic guidance for placement of fiducial markers into the pancreas will have the 19 gauge technique (ARM 1) of EUS guided fiducial marker technique.
  Interventions: Device: 19 Gauge EUS FNA BNX
- 22 Gauge EUS FNA BNX (Active Comparator): Subjects receiving EUS and fluoroscopic guidance for placement of fiducial markers into the pancreas will have the 22 gauge technique (ARM 2) of EUS guided fiducial marker technique.
  Interventions: Device: 22 Gauge EUS FNA BNX

INTERVENTIONS:
Device: 19 Gauge EUS FNA BNX — There will be fiducials placed in the pancreas according to facility policy and procedure utilizing the 19 gauge needle.
  Arms: 19 Gauge EUS FNA BNX
Device: 22 Gauge EUS FNA BNX — There will be fiducials placed in the pancreas according to facility policy and procedure utilizing the 22 gauge needle.
  Arms: 22 Gauge EUS FNA BNX

SUMMARY:
Comparison Study between 19 gauge EUS FNA BNX Needle vs. 22 gauge EUS FNA BNX Needle in Pancreatic Fiducial Placement To Treat Pancreatic Cancer

DETAILED DESCRIPTION:
A prospective multicenter study to compare the cost, time, complications, and migrations rate of two commercially available FDA approved needles; 19 gauge endoscopic ultrasound (EUS) fine needle aspiration (FNA) BNX needles to 22 gauge EUS FNA BNX needles.

There will be fiducials placed in the pancreas according to facility policy and procedure.

This is a randomized prospective multicenter trial. A minimum of 14 patients and a maximum of 30 patients will be enrolled at up to ten participating sites. Enrollment is projected to be complete within approximately one year.

Adult subjects with a diagnosis of pancreatic cancer who will receive SBRT for pancreatic cancer via Cyberknife or Tomotherapy will undergo EUS guided fiducial marker placement.

Subjects will be randomized to receive fiducial marker placement with either a 19 gauge EUS, FNA BNX needle or a 22 gauge EUS, FNA BNX needle. For all patients, standard hospital protocol will be followed for EUS procedures and patient care management.

The study duration will commence at the time of EUS guided fiducial marker placement and conclude at the time of last SBRT to the pancreas.

Cost effectiveness will be evaluated by providing an itemized statement, including anesthesiologist, and endoscopist charges. Time of procedure will be evaluated at time point of first lead needle loaded to time of last marker placed. Time measurement will begin when Endoscopist inserts the echoendoscope into the patient. Thus the patient is under anesthesia, in position, and staff is ready for the case. The time ends once last fiducial marker is placed. Complications will be reported and may include but not limited to pain, bleeding, peritonitis, and pancreatitis. Migration will be reported during the timeframe from simulation to the last day of SBRT.

The ability to receive SBRT from this EUS guided fiducial placement will be reported as simply a yes or no. Sites will provide a de-identified itemized statement for EUS guided fiducial placement procedure, prior to any discounted rate, including the endoscopist and anesthesiologist.

Follow up evaluations and treatment for pancreatic cancer will be performed in accordance with standard of care procedures and procedures deemed necessary by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects that plan to undergo CyberKnife treatment for pancreatic cancer
2. Subjects that are deemed physically able to undergo anesthesia (either Monitored Anesthesia Care (MAC) or general anesthesia)
3. Subjects (or the subjects Legally Authorized Representative [LAR]) that have agreed to participate in the study and have signed Informed Consent
4. Subjects 18 years of age or older
5. Subject must be able to hold anticoagulants as per institutional standard of care
6. Women of child bearing potential who are not pregnant as proven by a negative pregnancy test

Exclusion Criteria:

1. Subjects that are unable to tolerate anesthesia for the procedure
2. Subjects 17 or under
3. Subjects that refuse treatment for pancreatic cancer d Subjects whose anticoagulants cannot be held

e. Subjects who have distant metastatic disease f. Subjects who cannot or refuse EUS guided procedures. g Subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Total Cost Comparison | Duration of Fiducial Placement Procedure; approx 30 minutes
  Total cost of EUS guided fiducial placement in the pancreas to facilitate SBRT treatment of pancreatic cancer.
Total Time Comparison | Duration of fiducial placement procedure; up to 30 minutes
  Time comparison of EUS guided fiducial placement in the pancreas to facilitate SBRT treatment

SECONDARY OUTCOMES:
Migration Comparison | Duration of SBRT treatment; up to 8 weeks.
  The migration rate of pancreatic fiducials between placement and SBRT treatment
Complication Comparison | Duration of SBRT treatment; Up to 8 weeks
  Comparison of any fiducial related complications following placement

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sharma, MD, Principal Investigator — Parkview Health
Locations (1):
- Parkview Cancer Institute, Fort Wayne, Indiana, United States

DOCUMENTS (1):
  • Study Protocol (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT02376543/Prot_000.pdf